CLINICAL TRIAL: NCT02389257
Title: Optically Pumped 4He Magnetometers Performances Compared With Medical Reference Methods : Electrocardiography (ECG) and Magnetoencephalography (MEG)
Brief Title: Optically Pumped 4He Magnetometers Performances Compared With Medical Reference Methods (ECG and MEG)
Acronym: MINIMAG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MINIMAG
Record Dates: First submitted 2015-01-08; First posted 2015-03-17 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Magnetoencephalography; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MINIMAG / MEG (Experimental): Cerebral magnetic fields
  Interventions: Device: MINIMAG / MEG
- MINIMAG / ECG (Experimental): Cardiac magnetic fields
  Interventions: Device: MINIMAG / ECG

INTERVENTIONS:
Device: MINIMAG / MEG
  Arms: MINIMAG / MEG
Device: MINIMAG / ECG
  Arms: MINIMAG / ECG

SUMMARY:
Optically Pumped 4He Magnetometers operability for cerebral and cardiac magnetic fields measurement.

DETAILED DESCRIPTION:
Optically Pumped 4He Magnetometers vs reference sensors electrocardiogram (ECG) or SQUIDs data acquisitions

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old
* patient affiliated to social security or similarly regime
* informed consent form signed
* without cardiac, neurologic, psychiatric or metabolic medical history.

Exclusion Criteria:

* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Person with any implant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse EventsMagnetic brain or cardiac activity | 1 year
  Measure of Safety and Tolerability

SECONDARY OUTCOMES:
Brain or cardiac magnetic activity (Cerebral or cardiac magnetic fields record) | 1 hour
  Cerebral or cardiac magnetic fields record

CONTACTS AND LOCATIONS:
Locations (1):
- CLINATEC, Grenoble, France